CLINICAL TRIAL: NCT01816854
Title: Endovascular Treatment of Atherosclerotic Lesions in the SFA Using the Sinus-superflex-635 Stent
Status: Completed | Type: Observational
Sponsor: be Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BM-HERO-07-001
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Atherosclerotic Heart Disease
Keywords: Peripheral artery disease; SFA; PPA; Self-expandable nitinol stent; Endovascular; Stenosis; Primary pantency
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease; Constriction, Pathologic | interventions — Stents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with PAD
  Interventions: Device: Stenting

INTERVENTIONS:
Device: Stenting

SUMMARY:
In this prospective study, a newly developed self-expanding nitinol stent is evaluated for the treatment of atherosclerotic lesions in the superficial femoral artery and proximal popliteal artery.

ELIGIBILITY:
Inclusion Criteria:

* Patient must sign informed consent prior to the index-procedure
* Patient must be older than 18 years
* Patient must be compliant with follow-up dates at 1 month and 12 months
* Patients with intermittent claudication (Rutherford 2-3) and critical limb ischemia (Rutherford 4-5)
* Target lesion is located in the superficial femoral artery (minimal 1 cm from origin of SFA and minimal 1 cm above the edge of the patella)
* Reference vessel diameter ≥4.5 and ≤6.5 mm (visual estimate)
* Patients with a TASC A, B or C lesion
* Diameter stenosis of target lesion >50% or chronic occlusions
* Inflow arteries are free of hemodynamically significant obstruction (i.e. ≥50%)
* The popliteal artery (outflow) is free of hemodynamically significant obstruction (i.e. ≥50%)
* At least 1 patent below-the-knee vessel (anterior tibial artery, posterior tibial artery or peroneal artery) till the ankle confirmed by baseline angiography

Exclusion Criteria:

* Patients with Rutherford 1 and 6
* Patiens with Serum creatinine > 2.0 mg/dL or renal dialysis
* Patient takes esomeprazole or omeprazole
* Patient is pregnant
* Patient suffers from acute limb ischemia defined as any sudden decrease in limb perfusion causing a potential threat to limb viability
* Target lesion cannot be crossed with a guidewire
* Target lesion is located in the popliteal artery
* Patients with a nickel-titanium allergy
* Patients with an aneurysm in the superficial femoral artery and popliteal artery
* Patients with a TASC D lesion
* Patients with a life expectancy <1 year
* Patients with scheduled elective non-vascular procedures within 3 months after index-procedure, vascular procedures are allowed within 3 months after index-procedure if it is guaranteed that acetylic salicylic acid and clopidogrel intake is not interrupted
* Patients with previous bypass surgery in the SFA
* Patients with intolerance to antithrombotic medication (acetylic salicylic acid, clopidogrel, ticlopidine, glycoprotein IIb/IIIa inhibitors, direct thrombin inhibitors, etc)
* Patient has not been premedicated with acetylic salicylic acid (at least 80 mg/day) 2 hours before the index-procedure
* Patient has not been premedicated with clopidogrel (600 mg/day) 2 hours before the index-procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who suffer from intermittent claudication and critical limb ischemia (TASC A, B and C lesions).
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2012-10-08 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Binary restenosis | 12 months
  Binary restenosis is defined as a re-obstruction ≥ 50% of the target lesion (peak systolic velocity ratio > 2.4).

SECONDARY OUTCOMES:
Immediate procedural outcome (procedural, technical and device success) | peri-procedural
  Procedural success: combination of technical success, device success and absence of procedural complications.
  Technical success: successful vascular access and completion of the endovascular procedure and immediate morphological success with less than 30% residual diameter reduction of the treated lesion on completion angiography.
  Device success: exact deployment of the device according to the instructions for use as documented with suitable imaging modalities and in case of digital substraction angiography, in at least two different imaging projections.
Distribution of Rutherford stages | 12 months
Primary sustained clinical improvement | 12 months
  Defined as sustained upward shift of at least one category on the Rutherford classification without the need for repeated target lesion revascularization (TLR) in surviving patients.
Secondary sustained clinical improvement at 12 months | 12 months
  Defined as sustained upward shift of at least one category on the Rutherford classification including the need for repeated TLR in surviving patients.
Mortality | 30-day mortality
  post-procedural
Mortality | 12 months
Repeated target lesion revascularization (TLR) rate | 12 months
Repeated target extremity revascularization (TER) rate | 12 months
Amputation rate | 12 months
Rate of patient clopidogrel resistance | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Hendriks, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Antwerp, Belgium